CLINICAL TRIAL: NCT05036720
Title: Partner Inclusive Culturally Adapted Low-cost Group Parenting Programme for Depressed Fathers: A Cluster, Randomized Controlled Trial.
Brief Title: LTP Plus Dads-Partner Inclusive Intervention for Depressed Fathers in Pakistan
Acronym: LTP+Dads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: Grand Challenges Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LTP+Dads TTS-1
Record Dates: First submitted 2021-08-30; First posted 2021-09-08 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Depression
Keywords: Parenting Intervention; Partner Inclusive; Low and middle-income country; Paternal Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LTP+Dads (Experimental): Participants in this arm will be offered the LTP+Dads intervention. The intervention will be delivered by trained Community Health Workers (CHWs). This will be co-facilitated by LTP+ master trainers.
  Interventions: Behavioral: LTP+Dads
- Wait-list control: (Other): Participants in this arm will be offered the intervention once the LTP+ arm have completed their outcome assessment. For example, in each Union Council (UC) once the LTP+ arm has completed the intervention and 4th month outcome assessment the wait-list control group in the same UC will be offered the intervention.
  Interventions: Behavioral: LTP+Dads
- Optional mothers component (Other): To facilitate changes in co-parenting and optimize impact on child development, the partners of fathers who participate will be offered optional LTP+ group sessions running parallel to LTP+Dads.
  Interventions: Behavioral: LTP+ Optional mother component

INTERVENTIONS:
Behavioral: LTP+Dads — LTP+Dads is a 12 - session group integrated parenting intervention which includes a pictorial calendar, consisting of stages of child development from birth to 3 years. It includes parent-child play and other activities that promote parental involvement, learning, and attachment.
  The second component of the intervention is Cognitive Behaviour Therapy (CBT) adapted from the Jeanne Miranda manual (Group CBT for Depression) focusing on three areas: thoughts and your mood, activities and your mood, people interaction and your mood.
  The third component of intervention is content taken from Ed Bader's manual (Focus on Fathers) includes importance of fathers in child development, stress management at work and home, budgeting, anger management, conflict resolution and time management.
  Arms: LTP+Dads; Wait-list control:
Behavioral: LTP+ Optional mother component — LTP+ is comprised of two components; Learning through play (LTP) and Cognitive Behavior Therapy (CBT). The LTP+ is a low-literacy, sustainable program intended to provide parents with information on the healthy growth and development of their young children. The LTP research-based activities enhance children's development while simultaneously promoting attachment security through building parents' ability to read and be sensitive to their children's cues and through active involvement in their children's development. Plus the Thinking Healthy Program (THP) which adopts 'here and now' problem-solving approach. THP uses cognitive behavior therapy (CBT) techniques of active listening, changing negative thinking, and collaboration with the family.
  Arms: Optional mothers component

SUMMARY:
The aim of this study is to support and equip fathers and mothers with cognitive behavioral tools and knowledge about child development to be effective in their role as co-parent and partner, leading to improvement in paternal depression.

Objectives:

* To evaluate the clinical and cost effectiveness of the Learning Through Play+ (LTP + ) intervention in reducing depression in fathers and mothers.
* To evaluate the effectiveness of the LTP+ intervention in improving child outcomes.
* Process evaluation and identifying challenges in transition to scale up of the intervention across Karachi, Pakistan from the perspective of fathers, mothers, and other stakeholders.

DETAILED DESCRIPTION:
Parental depression is the leading cause of disability worldwide and low- and middle-income countries (LMIC) carry over 80% of this disease burden. Furthermore, parenting is a likely key mechanism for the intergenerational transmission of mental health risk particularly in LMICs as poverty undermines nurturing care in favour of survival. In LMICs, three quarters of young children experience physical discipline and harsh, coercive parenting is widespread. These issues are compounded by a lack of child and family policies. Attempts have been made to address maternal postnatal depression in LMICs, adopting parenting interventions mainly developed in high income countries (HIC) with improvements found in the home environment and maternal knowledge. The lack of focus on fathers may undermine intervention efforts to address depression in the current situation with Covid 19. Recognising the father as a key influencer in the family offers an alternative, systemic approach to breaking the intergenerational cycle of depression and fear during this pandemic, as well as directly addressing the father's own mental health. By alleviating paternal depression in the child's early years, a father is in a unique position to influence maternal wellbeing and his child's positive development. The novel aspect of the proposed project is the delivery of an innovative psychosocial intervention to depressed fathers. The fathers will receive a culturally adapted manual assisted group parenting intervention that incorporates a psychoeducational parenting programme i.e Learning Through Play (LTP) for fathers integrated with group cognitive behaviour therapy (CBT). Their partners (mothers) will be offered optional LTP+ developed for mothers. The study will be conducted in 18 towns across the city of Karachi, the largest city in Pakistan with a population of approximately 23 million. with Aa total of 2880 depressed fathers and their partners will participate in the study. In addition, a total of 4000 Community health workers(CHWs) will be trained in the LTP+ training program across Pakistan

ELIGIBILITY:
Inclusion Criteria:

* Fathers with a child aged 0-30 months
* We will also include those fathers who have partners in their third trimester of the pregnancy.
* All participants (fathers) over 18 years.
* All fathers with a diagnosis of major depressive disorder (using the Structured Clinical Interview for DSM-5)
* Ability to understand and complete the baseline assessment.
* If the pandemic continues, having access to any of the video calling services such as Skype/Zoom will be required. Fathers who do not have access to digital platforms will be provided smartphones throughout the trial period.

Exclusion Criteria:

* Any acute severe mental/physical illness or intellectual disability, which prevents fathers from participation.
* Active suicidal ideation
* Temporary residency indicating that they may be unlikely to be available for follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 2884 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HAM-D) (Hamilton, 1960) | Changes from baseline to 4th and 6th month
  This is the most widely used clinician-rated depressive symptom scale, is validated in Urdu, and was used in our exploratory LTP Plus Dads trial. Higher score indicates more severe depression. Minimum score is 0 and maximum score is 68

SECONDARY OUTCOMES:
Structured Clinical Interview for DSM-5 (SCID) (Spitzer, Williams, Gibbon, & First, 1992): | Baseline
  The SCID is a semi-structured diagnostic interview which has been widely used in cross-national epidemiological and treatment studies (Weissman et al., 1996). The interview consists of standardized diagnostic questions arranged in modules corresponding to each DSM-V disorder. This interview will be conducted by trained psychologists.
Patient Health Questionnaire (PHQ-9) (Löwe, Kroenke, Herzog, & Gräfe, 2004): | Changes from baseline to 4th and 6th month
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. Higher score indicates more severe depression. Scores ranging from 1-4 Minimal depression, 5-9 Mild depression,10-14 Moderate depression,15-19 Moderately severe depression, 20-27 Severe depression.
Generalised Anxiety Disorder Assessment (GAD-7) (Spitzer, Kroenke, Williams, & Löwe, 2006): | Changes from baseline to 4th and 6th month
  A 7-item scale measuring generalised anxiety. GAD-7 total score for the seven items ranges from 0 to 21. Higher score indicates more severe anxiety.
Parenting Stress Index (PSI -Short Form) (Haskett, Ahern, Ward, & Allaire, 2006): | Changes from baseline to 4th and 6th month
  A 36-item perceived stress measure in 3 subscales, parenting distress, difficult child characteristics, and dysfunctional parent-child interaction. A Total score is calculated by summing the three subscales scores, ranging from 36 to 180. Scores of 90 or above may indicate a clinical level of stress. Higher score indicates more severe parenting stress.
How Are You Feeling (Andrew Haig., 2008) | Changes from baseline to 4th and 6th month
  This picture booklet can help the early detection of mood disturbance in pregnancy and/or following childbirth. The booklet can be used by a verity of health workers or support workers. It is designed to assess the feelings today and in the past few days and to talk about moods, emotions and general health." Higher score indicates more severe depression
Knowledge, Attitudes and Practices (KAP) (Rahman et al., 2009): | Changes from baseline to 4th and 6th month
  A 25 -item questionnaire of paternal knowledge and expectations for child development in the first three years. Higher score indicate (ranging from 0 to 25) better knowledge about child development.
Hurt, Insulted, Threatened with Harm and Screamed (HITS) (Sherin, Sinacore, Li, Zitter, & Shakil, 1998) | Changes from baseline to 4th and 6th month
  A 4-item intimate partner violence screener producing a score of 4-20. Higher score indicates more severe level of violence
Euro-Qol Five- Dimensions (EQ-5D-5L) (Herdman et al., 2011): | Changes from baseline to 4th and 6th month
  Health-related quality of life as measured for mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems. In addition, there is a visual analogue scale (VAS) to indicate the general health status with 100 indicating the best health status.
Client Service Receipt Inventory (CSRI) (Beecham & Knapp, 1995): | Changes from baseline to 4th and 6th month
  It is used to collect information on the whole range of services and supports study participants may use. This data can be used for a wide range of applications, including estimating the costs of service receipt.
Dyadic Adjustment Scale(DAS):(Spanier, 1976) | Changes from baseline to 4th and 6th month
  DAS is a 32 items self-report questionnaire, to measure couple satisfaction and to assess how each partner perceives his/her relationship. The scale has good psychometric properties (Graham, Liu, & Jeziorski, 2006) and has also been used with depressed mothers (Wolman, Chalmers, Hofmeyr, & Nikodem, 1993). The resultant score ranges from 0 to 151, with higher scores indicating a more positive dyadic adjustment and a lower level of distress.
The Prodromal Questionnaire-(PQ-16) (Loewy, Bearden, Johnson, Raine, & Cannon, 2005): | Changes from baseline to 4th and 6th month
  A brief self-report screening questionnaire that assesses the presence of attenuated psychotic symptoms, the PQ-16 is a reliable measure and correlates well with the CAARMS. The scale has been used in a previous study in Pakistan (Qurashi et al., 2017). Higher score (range 0-16) indicates more probability of having psychosis.
World Health Organization Disability Assessment Schedule 2.0 (World Health Organization, 2000) | Changes from baseline to 4th and 6th month
  The adult self-administered version of the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) is a 36-item measure that assesses disability in adults age 18 years and older. It assesses disability across six domains, including understanding and communicating, getting around, self-care, getting along with people, life activities (i.e., household, work, and/or school activities), and participation in society. Translated version of scale has been used in previous trials in Pakistan(Naeem et al., 2015) . Higher score indicates more disability, ranging from 0 to 100, where 0 = no disability; 100 = full disability.
Problem Solving Inventory-(PSI) (Heppner, 1988): | Changes from baseline to 4th and 6th month
  The PSI is one of the most widely used self-report inventories in problem solving. The PSI assesses an individual's awareness and evaluation of his or her problem-solving abilities or style, and this provides a global appraisal of that individual as a problem solver. Higher score indicates better problem solving that ranges from 32 to 192.
The General Self-Efficacy Scale (GSES) (Schwarzer & Jerusalem, 2010): | Baseline, 4th and 6th month
  The GSES is a simple 10 item self-administered scale. The scale is developed to assess a general sense of perceived self-efficacy with the aim to predict coping with daily hassles as well as adaptation after experiencing all kinds of stressful life events. A total score ranges from 10 to 40. Higher scores indicate higher perceived general self-efficacy, lower scores indicate lower perceived general self-efficacy.
The Postpartum Bonding Questionnaire (PBQ) (Brockington, Fraser, & Wilson, 2006): | Changes from baseline to 4th and 6th month
  The PBQ is designed to detect disturbance in the mother-child relationship. The scale has25 items, each followed by six alternative responses ranging from 'always' to 'never'. Positive responses, such as ''I enjoy playing with my baby'', are scored from zero ('always') to 5 ('never'). Negative responses, such as ''I am afraid of my baby'', are scored from 5 ('always') to zero ('never'). A high score indicates pathology in mother-child relationship. Higher score indicates more strong bonding
Assessment of the growth and development of children: Weight | Change in weight from Baseline and 6th month
  Data on child growth: Anthropometric measures of child growth will be collected through measuring children's weight in kilogram
Assessment of the growth and development of children: Height | change in height from Baseline and 6th month
  Data on child growth: Anthropometric measures of child growth will be collected through measuring children's height in meters at baseline, and 6 months after baseline.
Assessment of the growth and development of children: Head circumference | change in head circumference measurement from Baseline and 6th month
  Data on child growth: Anthropometric measures of child growth will be collected through measuring children's head circumference in centimeters at baseline, and 6 months after baseline.
Ages and Stages Questionnaire (ASQ) and ASQ Socio-emotional Scales (ASQ: SE) (Squires et al., 2015), | Changes from baseline to 4th and 6th month
  parent-reported screening instrument comprising of 25/29 items on social and emotional difficulties recommended for evaluating early interventions.
Manchester Assessment of Caregiver-Infant Interaction (MACI) (Wan, Brooks, Green, Abel, & Elmadih, 2017): | Baseline and 4th month
  This validated global rating measure evaluates qualities of observed parent-child interaction from 6-minute video clips of unstructured play interaction. It comprises of seven seven-point rating scales that covers key characteristics of interaction, such as caregiver sensitive responsiveness, child attentiveness to caregiver, and level of mutuality, which are understood to reflect the quality of the parent-child relationship and the child's social and emotional environment. Due to the resource requirements of an observational measure, 5% from each intervention arm will be selected randomly for MACI assessment.
Bayley Scales of Infant Development (Bayley, 1993): | Baseline and 6th month
  It is a standard series of measurements to assess the development of infants and toddlers, ages 1-42 months. This measure consists of a series of developmental play tasks and takes between 45 - 60 minutes to administer. The Bayley is an early childhood, norm-referenced assessment instrument that evaluates the current level of functioning for young children. The instrument, which is individually administered by qualified professionals, assesses developmental domains such as language, cognitive, personal/social, fine motor, and gross motor skills. The assessment of these skills in conjunction with other forms. Other specific purposes of the Bayley are to identify possible developmental delays and inform professionals about specific areas of strength or weakness when planning a comprehensive intervention and provide a method of monitoring a child's developmental progress.
Home Observation for Measurement of the Environment (HOME) (Caldwell & Bradley, 1984): | Changes from baseline to 4th and 6th month
  HOME is a descriptive proﬁle which yields a systematic assessment of the caring environment in which the child is reared. The primary goal of the scale is to measure, with in a naturalistic context, the quality and quantity of stimulation and support available to a child in home environment. It contains 45 items under 6 subscales which are; 1. Emotional and verbal responsively of the primary caregiver (item 1-11); 2. Avoidance of restriction and punishment (item 12-19); 3. Organization of the physical and temporal environment (item 20-25); 4. Provision of appropriate play materials (item 26-34); 5. Parental involvement with the child (item 35-40), 6. Opportunity for variety in daily stimulation (item 40-45).
World Health Organisation Quality of Life (WHOQOL-BREF) (WHO, 1997) | Changes from baseline to 4th and 6th month
  The WHOQOL-BREF is a self-administered questionnaire comprising 26 questions on the individual's perceptions of their health and well-being over the previous two weeks. Responses to questions are on a 1-5 Likert scale where 1 represents "disagree" or "not at all" and 5 represents "completely agree" or "extremely.

OTHER OUTCOMES:
Kessler Psychological Distress Scale (K10) (Andrews & Slade, 2001): | Changes from baseline to 4th month
  It is used to measure psychological distress. It's a 10-item scale measuring emotional states with a 5-level response scale. We will use this measure with community health workers before and after training. Higher score indicates more severe stress, ranging from 10- 50.
The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): | Changes from baseline to 4th month
  we will be using the Short Warwick Edinburgh Mental Wellbeing 7 items Scale (SWEMWBS) (Tennant et al., 2007), where a higher score indicates greater psychological wellbeing. Administration time: 3-6 minutes. We will use this measure with community health workers before and after training.
Weiman Occupational Stress Scale:(Weiman, 1978): | Changes from baseline to 4th month
  Job related stress will be measured using Weiman Occupational Stress scale. We will use this measure with community health workers before and after training.

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Chaudhry, MD, Principal Investigator — Pakistan Institute of Living and Learning; Muhammad Ishrat Husain, MD, Principal Investigator — Centre for Addiction and Mental Health,Canada
Locations (1):
- 18 Towns, Karachi, Sindh, Pakistan